CLINICAL TRIAL: NCT01941810
Title: A Pilot Study of Bovine Lactoferrin in Cancer Patients Reporting Taste Disturbances While Receiving Chemotherapy
Brief Title: Bovine Lactoferrin Supplement in Improving Taste in Patients With Cancer Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00025192; NCI-2013-01741 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98513 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Anorexia; Cachexia; Malignant Neoplasm; Oral Complications of Chemotherapy
MeSH Terms: conditions — Anorexia; Cachexia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (bovine lactoferrin supplement) (Experimental): Patients receive bovine lactoferrin supplement PO TID for 1 month.
  Interventions: Dietary Supplement: bovine lactoferrin supplement; Other: questionnaire administration; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: bovine lactoferrin supplement — Given PO
  Other Names: bLF supplement
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies how well bovine lactoferrin supplement works in improving taste in patients with cancer receiving chemotherapy. Bovine lactoferrin supplement may help improve the ability to taste food in patients who are receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the impact of lactoferrin supplementation (bovine lactoferrin supplement) on self-reported taste and smell disturbances in cancer patients receiving chemotherapy.

SECONDARY OBJECTIVES:

I. To assess the impact of lactoferrin supplementation on the baseline lipid peroxidation byproducts in saliva in cancer patients as measured by the thiobarbituric acid reactive substances (TBARs) assay.

II. To assess the impact of lactoferrin supplementation on the ability of cancer patients to generate increased lipid peroxidation byproducts when challenged with a weak iron-containing solution.

III. To assess the impact of lactoferrin supplementation on self-reported general quality of life and on specific self-reported anorexia/cachexia issues in cancer patients with established chemotherapy-induced taste disturbances.

IV. To assess the incidence of vitamin D deficiency in cancer patients with chemotherapy induced taste changes.

OUTLINE:

Patients receive bovine lactoferrin supplement orally (PO) three times daily (TID) for 1 month.

After completion of study treatment, patients are followed up at 2 weeks and 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed carcinoma of any site; the two exceptions are pancreatic cancer and colon cancer patients who are receiving oxaliplatin; those patients will be ineligible for participation in this current study but will be eligible for Comprehensive Cancer Center of Wake Forest University (CCCWFU) 98112 instead
* There are no restrictions on the amount or types of prior therapy; eligible patients must be receiving ongoing chemotherapy that is planned to continue for at least one month following enrollment in this trial; any dose or schedule of chemotherapy administration is allowed as long as patients have self-reported taste disturbance that has either: 1) developed since the initiation of chemotherapy, or 2) a pre-existing, treatment-induced taste disturbance has subjectively worsened since initiating chemotherapy
* Patients must have normal baseline self-reported taste perception prior to the development of cancer
* Life expectancy of >= 3 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with a subjective history of an extreme dry mouth syndrome that prevents them from producing adequate amounts of saliva (approximately 2 mL in 15-20 min)
* Patients known to be human immunodeficiency virus (HIV)-positive
* Patients with any of the following conditions: untreated gastrointestinal reflux disease; untreated diabetes mellitus; active thrush; active oral infection; active mucositis
* Patients who are pregnant or breastfeeding are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in taste disturbances using the visual analogue scale (VAS) and the Smell and Taste Questionnaire | Baseline to up to 1 month
  Tested separately by using paired t-tests to assess the significance of the baseline to one month changes.
Change in smell disturbances using the VAS and the Smell and Taste Questionnaire | Baseline to up to 1 month
  Tested separately by using paired t-tests to assess the significance of the baseline to one month changes.

SECONDARY OUTCOMES:
Effect of bovine lactoferrin supplement on lipid peroxidation byproducts as measured by the TBARs assay | Up to 2 months
Malondialdehyde (MDA) concentrations before and after a ferrous iron oral rinse | Up to 2 months
Smelling loss as quantified by the Brief Smell Identification Test (B-SIT) | Up to 2 months
Quality of life as quantified by the Functional Assessment of Anorexia/Cachexia Treatment (FAACT) and Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) questionnaires | Up to 2 months

OTHER OUTCOMES:
Proportion of patients with vitamin D deficiency | Baseline
  The estimated proportion deficient will be calculated as the number deficient divided by the total number of patients. An exact binomial 95% confidence interval will be calculated for this estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Virginia Polytechnic Institute and State University, Blacksburg, Virginia